CLINICAL TRIAL: NCT00277238
Title: CPG 10101 Combination Therapy for the Treatment of Hepatitis C: A Phase II Randomized, Open Label, Multi-Center, Parallel Arm, Controlled Trial of CPG 10101 at Two Different Dose Levels With Pegylated-Interferon-Alpha 2B (PEG-IFN) Plus Ribavirin (RBV) or PEG-IFN Plus RBV Without CPG 10101 in the Treatment of Non-Responder (Null and Partial Responder) HCV Genotype 1 Infected Subjects
Brief Title: CPG10101 Combination Therapy For The Treatment Of Hepatitis C In Non-Responder (Null And Partial Responder) Hepatitis C Virus (HCV) Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1211002; CPG 10101-004
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis, Chronic Active
Keywords: HCV; Hepatitis c virus; Virus diseases; Interferon-alpha; Interferons; Liver diseases
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C; Virus Diseases; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CPG10101 (0.2) + pegylated inteferon + ribavirin (Experimental)
  Interventions: Drug: CPG10101
- CPG10101 (0.5) + pegylated inteferon + ribavirin (Experimental)
  Interventions: Drug: CPG10101
- Pegylated interferon + ribavirin (Active Comparator)
  Interventions: Drug: Control
- CPG10101 + pegylated interferon + ribavirin (rollover) (Experimental)
  Interventions: Drug: CPG10101

INTERVENTIONS:
Drug: CPG10101 — CPG10101, subcutaneous, 0.2mg/kg, weekly, 24wks Pegylated interferon alfa-2b, subcutaneous, 1.5ug/kg, weekly, 24wks Ribavirin, oral, 800-1400mg/day (weight-based), daily, 24wks
  Arms: CPG10101 (0.2) + pegylated inteferon + ribavirin
Drug: CPG10101 — CPG10101, subcutaneous, 0.5mg/kg, weekly, 24wks Pegylated interferon alfa-2b, subcutaneous, 1.5 ug/kg, weekly, 24wks Ribavirin, oral, 800-1400mg/day (weight-based), daily, 24wks
  Arms: CPG10101 (0.5) + pegylated inteferon + ribavirin
Drug: Control — Pegylated interferon alfa-2b, subcutaneous, 1.5 ug/kg, weekly, 12wks Ribavirin, oral, 800-1400mg/day (weight-based), daily, 12wks
  Arms: Pegylated interferon + ribavirin
Drug: CPG10101 — CPG10101, subcutaneous, 0.5mg/kg, weekly, 24wks Pegylated interferon alfa-2b, subcutaneous, 1.5 ug/kg, weekly, 24wks Ribavirin, oral, 800-1400mg/day (weight-based), daily, 24wks
  Arms: CPG10101 + pegylated interferon + ribavirin (rollover)

SUMMARY:
The purpose of this study is to determine the efficacy and tolerability of CPG 10101 at two different dose levels with pegylated-interferon-alpha 2B (PEG-IFN) plus ribavirin (RBV) compared to PEG-IFN and RBV without CPG 10101 in HCV positive subjects who were classified as non-responders to previous adequate PEG-IFN plus RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

HCV positive subjects documented by serum HCV RNA concentration > 100,000 IU/mL within 21 days of first study treatment Receipt of adequate previous PEG-IFN and RBV therapy for a minimum of 12 weeks (PEG-IFN alpha-2a doses of > 180 μg/wk or PEG-IFN alpha-2b 1.5 µg/kg/wk and at least 800 mg RBV daily) not resulting in a minimum of a 2 log decrease in HCV RNA concentrations while on treatment (null responders). Or, receipt of adequate previous treatment PEG-IFN and RBV therapy for a minimum of 24 weeks (PEG-IFN alpha-2a doses of ≥ 180 μg/wk or PEG-IFN alpha-2b 1.5 µg/kg/wk and at least 800 mg RBV daily) resulting in a minimum of a 2 log decrease in serum HCV RNA concentrations by 12 weeks of treatment but not resulting in an undetectable viral load after 24 weeks of treatment (partial responders). If dose modifications were necessary during the treatment due to adverse events, the subject must have received at least 80% of the PEG-IFN dose and 80% of the RBV dose to be eligible for the study.

HCV genotype 1 only; other HCV genotypes are excluded. Adults, 18+ years old Written informed consent Liver biopsy within 5 years of the first dose of study drug, documenting changes consistent with hepatitis C

Adequate bone marrow, liver, and renal function demonstrated by:

* Hemoglobin > 12 g/dL for females and > 13 g/dL for males
* White blood cell (WBC) > 3,000/mm3
* Neutrophils > 1,500/mm3
* Platelets > 80,000/mm3
* Total bilirubin < 1.6 mg/dL
* Direct bilirubin < 1.5 upper limit of normal. If indirect bilirubin is elevated, Gilbert's disease must be documented in chart and substantiated.
* Albumin > 3.7 g/dL and < 4.9 g/dL
* Serum creatinine < upper limit of normal per central laboratory. If serum creatinine is > upper limit of normal then calculated creatinine clearance has to be > 100 mL/min (by Cockcroft-Gault formula) for patient to be eligible.

Negative pregnancy test in women of childbearing potential. Females of childbearing potential and males who have partners of childbearing potential must use two forms of effective contraception during treatment and during the 6 months after treatment has been concluded.

Serum thyroid stimulating hormone (TSH) levels within normal ranges within 21 days of first study treatment, regardless of treatment with L-thyroxin.

Exclusion Criteria:

Treatment with any IFN based therapies and/or antiviral therapies within 30 days of the first dose of study drug Subjects who have previously received an HCV vaccine Child-Pugh Class B or C History of psychiatric conditions including, but not limited to, psychosis, suicidal ideations, or major depression. Subjects with mild to moderate depression in the past who have a normal to mild Beck Depression Inventory score and no prior history of suicidal gestures or attempts may be enrolled if, in the Investigator's opinion, they are suitable for treatment.

Significant cardiovascular disease (e.g., New York Heart Association [NYHA] class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; or uncontrolled atrial or ventricular cardiac arrhythmias) History of immunodeficiency or autoimmune disease including autoimmune hepatitis, allogeneic transplant, or pre-existing autoimmune or antibody-mediated disease including, but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.

Other serious medical conditions including, but not limited to:

* HIV-1
* Hepatitis B (positive hepatitis B surface antigen [HBsAg])
* Cancer (active tumors in the last 5 years)
* Pregnant, partners of pregnant women, or nursing women
* Alcohol or drug misuse within 90 days of screening Use of immunosuppressive doses of steroids or any anti-metabolite therapies within 3 months of entry into the study (inhaled and topical corticosteroids are permitted).

Receipt of any vaccine or immunoglobulin within 30 days before the first dose of study drug. Flu vaccines are only allowed once the subjects are qualified for 36 additional weeks of treatment.

Prior administration of oligodeoxynucleotides (including study medication CPG 10101), ribozymes, or any known allergy to CPG 10101, interferon, RVN or their excipients.

Receipt of any investigational drug therapy within 30 days before the first dose of study drug.

Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Serum HCV RNA concentrations, over 12wks, relative to baseline, early virologic response (EVR) | 12wks
Serum HCV RNA concentrations, 6months after treatment completed, relative to baseline, sustained virologic response (SVR) | 72wks

SECONDARY OUTCOMES:
Safety and Tolerability: adverse events, vital signs, clinical and laboratory parameters, depression score, physical exam, electrocardiogram (ECG), ophthalmologic exam (if required) | 28wks
Dose exposure | 24wks
Child-Pugh score | 24wks
Serum Biomarkers: cytokines and chemokines, over time, relative to baseline | 24wks
Immunophenotyping profile, over time, relative to baseline, HCV specific immune response, over time, relative to baseline, level of innate immune activation at baseline | 24wks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia